CLINICAL TRIAL: NCT02294344
Title: A Prospective, Controlled Study of Double Filtration Plasmapheresis (DFPP) in Patients With Antineutrophil Cytoplasmic Autoantibody Associated Glomerulonephritis (AAGN)
Brief Title: The Clinical Efficacy of DFPP in Patients With AAGN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of subject is very difficult.
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., Professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT1403
Record Dates: First submitted 2014-06-03; First posted 2014-11-19 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: double filtration plasmapheresis; ANCA-Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DFPP&CTX (Experimental): double filtration plasmapheresis(DFPP) combined with intravenous cyclophosphamide (IV-CTX) pulse therapy in addition(DFPP&CTX)
  Interventions: Other: DFPP&CTX
- cyclophosphamide (Active Comparator): cyclophosphamide(CTX) pulse therapy
  Interventions: Drug: CTX

INTERVENTIONS:
Other: DFPP&CTX — First,patients received methylprednisolone pulse therapy followed by oral prednisone and intravenous cyclophosphamide (IV-CTX) pulse therapy.
  Then double volume of plasma was processed during each DFPP session every two day. A fraction plasma separator(Asahi Kasei Medical, surface area 2.0 m2,pore size 0.03 mm)and another fraction plasma separator (Asahi Kasei Medical, surface area 2.0 m2, pore size 0.01 mm)were used as first and second filter for plasma fractionation, respectively. 1.5 volume of plasma was processed, and 35~45g human albumin and blood plasma was supplemented during each session. The patients were treated with DFPP every two days for at least 3 times. After DFPP, 300-500ml blood plasma was supplemented.
  Other Names: Double Filtration Plasmapheresis +cyclophosphamide
  Arms: DFPP&CTX
Drug: CTX — First,patients received methylprednisolone pulse therapy followed by oral prednisone and intravenous cyclophosphamide (IV-CTX) pulse therapy.
  After three months therapy, if the renal function was not recover, the patient would be withdrawn from the study. The other patients after CTX pulse therapy for 6 months and achieve remission to receive oral maintenance therapy with azathioprine (AZA).
  The dosage of AZA was 1.0-2.0mg/kg/d(more than 50mg/d) and adjusted by white cell count and liver enzyme. If white cell count <3×109/L or an increase in liver enzyme to more than twice the normal upper limit, the dosage of AZA should be reduced. If white cell count <3×109/L or liver enzyme increased repeatedly, the patient would be withdrawn from the study.
  Other Names: cyclophosphamide
  Arms: cyclophosphamide

SUMMARY:
The clinical efficacy of double filtration plasmapheresis(DFPP) in patients with antineutrophil cytoplasmic autoantibody associated glomerulonephritis(AAGN).

DETAILED DESCRIPTION:
This is a single center, prospective, randomized,controlled study to compare the clinical efficacy of double filtration plasmapheresis (DFPP) combined with intravenous cyclophosphamide (IV-CTX) pulse therapy versus IV-CTX pulse therapy in patients with antineutrophil cytoplasmic autoantibody associated glomerulonephritis(AAGN).

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ANCA associated vasculitis(AAV), using criteria adapted from the disease definitions of the Chapel Hill consensus conference
* serum positive ANCA and the ANCA level ≥100 relative unit/ml
* with renal involvement and serum creatinine≥3 mg/dl
* written informed consent had been provided.

Exclusion Criteria:

* other secondary vasculitis
* anti-glomerular basement membrane(GBM) positive
* severe infection; hepatitis B antigenemia, anti- hepatitis C virus
* immunodeficiency; or immunoglobulin G(IgG)<2g/l
* life threatening
* renal biopsy show globally sclerotic glomeruli>60% and normal glomeruli<10%
* need renal replacement therapy for more than 4w
* received large dose of methylprednisolone(MP),CTX,mycophenolate mofetil(MMF), plasmapheresis or intravenous immunoglobulin(IVIg) therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
the renal recovery rate | 3 months
  the renal recovery rate at 3 mo defined by dialysis independence and the SCr <5mg/dl for the patients needed renal replacement therapy at the basement, or the SCr decreased more than 30% of the baseline and the urine sediment red blood cell less than 50*104/ml for the patients without renal replacement at the basement.

SECONDARY OUTCOMES:
kidney survival | 12 months
  patient and kidney survival at 12 month

OTHER OUTCOMES:
the antineutrophil cytoplasmic antibodies(ANCA) level at 12 month | 12 months
relapse defined by birmingham vasculitis activity score(BVAS) increased more than 1.0 at 12 month | 12 months
the change of BVAS | 12 months
the change of Urine protein | 12 months
the change of the count of urine sediment red blood cell | 12 months
the change of the count of serum creatinine(SCr ) | 12 months
the change of estimated glomerular filtration rate(eGFR) | 12 months
the vasculitis damage index(VDI) at 12 month | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China